CLINICAL TRIAL: NCT00304512
Title: A Phase 2, Open-Label, Multiple Dose Level, 12-Week Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AT1001 in Female Patients With Fabry Disease
Brief Title: A 12-Week Safety and Pharmacodynamic Study of AT1001 (Migalastat Hydrochloride) in Female Participants With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAB-CL-204
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Substrate
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Migalastat Low Dose 50 mg (Experimental): Migalastat 50 mg was administered orally QOD during the 12-week treatment period and then during the optional 36-week treatment extension period.
  Interventions: Drug: migalastat HCl
- Migalastat Middle Dose 150 mg (Experimental): Migalastat 150 mg was administered orally QOD during the 12-week treatment period and then during the optional 36-week treatment extension period.
  Interventions: Drug: migalastat HCl
- Migalastat High Dose 250 mg (Experimental): Migalastat 250 mg was administered orally QOD during the 12-week treatment period and then during the optional 36-week treatment extension period.
  Interventions: Drug: migalastat HCl

INTERVENTIONS:
Drug: migalastat HCl
  Other Names: AT1001; Galafold; migalastat

SUMMARY:
Study to evaluate the safety, tolerability, and pharmacodynamics of migalastat hydrochloride (HCl) (migalastat) in participants with Fabry disease.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in female participants with Fabry disease. The study consisted of a 4-week screening period, during which participants' galactosidase (GLA) genotype was assessed for α-galactosidase A (α-Gal A) activity in response to migalastat. Participants were required to have α-Gal A activity responsive to migalastat. The study consisted of a 12-week treatment period, followed by an optional 36-week extension period. Participants received migalastat once every other day (QOD) for 12 weeks during the treatment period and the optional 36-week extension period for a total treatment duration of up to 48 weeks. Participants were stratified by α-Gal A enzyme activity (high >40%, and low ≤40%) then randomly assigned to receive migalastat at 1 of 3 specified dose levels (50, 150, or 250 milligrams [mg]).

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 65 years of age (inclusive)
* Heterozygous for Fabry disease
* Had a confirmed diagnosis of Fabry disease with a documented missense gene mutation (individual or familial)
* Had enhanceable enzyme activity based on in vitro tests
* Were naïve to enzyme replacement therapy (ERT) and other therapies, except for palliative therapies for the signs and symptoms of Fabry disease, or stopped ERT for at least 18 weeks
* Had end organ dysfunction, even minimal, demonstrated by abnormal electrocardiogram (ECG) or evidence of left ventricular hypertrophy documented by echocardiogram or by cardiac biopsy; or renal insufficiency documented by common clinical assessments such as creatinine and glomerular filtration rate or by renal biopsy; or brain tissue dysfunction as documented by evidence of stroke (clinically or imaging); or peripheral nervous tissue dysfunction documented by complaints of intolerance to heat or cold, decreased vibratory sense and proprioception, decreased ability to perspire, or acroparesthesia.
* Were willing to undergo 2 renal and 3 skin biopsies
* Agreed to be sexually abstinent or practice an effective method of contraception when engaging in sexual activity during the course of the study and for a period of 30 days following their completion of the study for women of childbearing potential.
* Were willing and able to provide written informed consent

Exclusion Criteria:

* Pregnant or lactating
* History of organ transplant
* History of significant disease other than Fabry disease (for example, end-stage renal disease; Class III or IV heart disease [per the New York Heart Association classification]; current diagnosis of cancer, except for basal cell carcinoma of the skin; diabetes [unless hemoglobin A1c ≤8]; or neurological disease that would have impaired the participant's ability to participate in the study)
* Serum creatinine >176 micromoles/liter on Day -2
* Screening 12-lead ECG demonstrating corrected QT interval >450 milliseconds
* Pacemaker or other contraindication for magnetic resonance imaging scanning
* Taking a medication prohibited by the protocol: Fabrazyme® (agalsidase beta), Replagal™ (agalsidase alfa), Glyset® (miglitol), Zavesca® (miglustat), or any experimental therapy for any indication
* Participated in a previous clinical trial in the last 30 days
* Any other condition which, in the opinion of the investigator would jeopardize the safety of the participant or impact the validity of the study results.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09-07 (Actual); Primary Completion 2008-05-09 (Actual); Study Completion 2008-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (6):
- Decatur, Georgia, United States
- Parkville, Victoria, Australia
- Porto Alegre, Brazil
- Montreal, Canada
- Paris, France
- Salford, United Kingdom

REFERENCES:
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681
- [Derived] Giugliani R, Waldek S, Germain DP, Nicholls K, Bichet DG, Simosky JK, Bragat AC, Castelli JP, Benjamin ER, Boudes PF. A Phase 2 study of migalastat hydrochloride in females with Fabry disease: selection of population, safety and pharmacodynamic effects. Mol Genet Metab. 2013 May;109(1):86-92. doi: 10.1016/j.ymgme.2013.01.009. Epub 2013 Jan 26. PMID 23474038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before randomization, participants were stratified into 2 groups (high or low) by their baseline α-galactosidase A (α-Gal A) activity. High was defined as activity greater than 40% of normal; low was defined as activity less than or equal to 40% of normal.
Groups:
- Migalastat Low Dose 50 mg: Migalastat 50 milligrams (mg) was administered orally QOD during the 12-week treatment period and then during the optional 36-week treatment extension period.
Period: Treatment Period
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Started | 2 | 4 | 3
Safety Population (Received at least 1 dose of study drug) | 2 | 4 | 3
Pharmacokinetic (PK) Population (Received study drug and had at least 1 postbaseline PK parameter recorded) | 2 | 4 | 3
Pharmacodynamic (PD) Population (Received study drug and had at least 1 postbaseline PD parameter recorded) | 2 | 4 | 3
Completed | 2 | 4 | 3
Not Completed | 0 | 0 | 0
Period: Extension Period
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Started | 2 | 4 | 3
Completed | 2 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg | Total
Number analyzed (Participants) | 2 | 4 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (18.38) | 44.8 (9.95) | 44.0 (2.65) | 45.4 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe adverse event was defined as an adverse event that was incapacitating and required medical intervention. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through Week 48 is presented. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Week 48
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Number analyzed (Participants) | 2 | 4 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: PK: Area Under The Concentration Versus Time Curve (AUC) After Administration Of Migalastat
Description: The AUC to the last measurable concentration (AUC0-t) was evaluated in plasma following a single oral dose of migalastat on Day 1 and following multiple oral doses on Day 14 (2 weeks) and Day 84 (12 weeks). All samples were collected on each dosing day.
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, and 10 hours (postdose)
Population: PK Population: all participants who received study drug and had at least 1 postbaseline PK parameter recorded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliters (ng*hr/mL)
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Number analyzed (Participants) | 2 | 4 | 3
nanograms*hours/milliliters (ng*hr/mL)
  AUC0-t: Single Dose, Day 1 | 2628.9 (100.4) | 8941.6 (32.2) | 13217.2 (30.2)
  AUC0-t: Multiple Dose, Day 14 | 3191.6 (64.9) | 10637.9 (35.6) | 14850.6 (9.6)
  AUC0-t: Multiple Dose, Day 84 | 2300.3 (79.6) | 8581.9 (29.7) | 9970.3 (37.8)

3. Secondary Outcome: α-Gal A Activity In Leukocytes At Baseline, Week 12, And Week 48
Description: Leukocytes were isolated from whole blood and lysed, and α-Gal A activity was measured using a validated fluorometric assay, with catalysis to fluorescent 4-methylumbelliferone (4-MU) as the activity measure. The activity values obtained were normalized to protein (measured using a colorimetric assay) and reported as enzyme activity (nanomole [nmol] 4-MU/hr) per mg of protein. On Day 1 of the first visit and at every visit thereafter, the samples were collected prior to dosing with migalastat. α-Gal A activity in leukocytes are presented by individual participants.
Time Frame: Baseline, Week 12 (end of treatment period), Week 48 (end of extension period)
Population: PD Population: all participants who received study drug and had at least 1 postbaseline PD parameter recorded.
Measure: Number; unit: nmol 4-MU/hr/mg protein
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Number analyzed (Participants) | 2 | 4 | 3
nmol 4-MU/hr/mg protein
  Participant 1: Baseline: number analyzed (Participants) | 1 | 0 | 0
  Participant 1: Baseline | 13.4 |  |
  Participant 1: Week 12: number analyzed (Participants) | 1 | 0 | 0
  Participant 1: Week 12 | 2.46 |  |
  Participant 1: Week 48: number analyzed (Participants) | 1 | 0 | 0
  Participant 1: Week 48 | 26 |  |
  Participant 2: Baseline: number analyzed (Participants) | 1 | 0 | 0
  Participant 2: Baseline | 24.5 |  |
  Participant 2: Week 12: number analyzed (Participants) | 1 | 0 | 0
  Participant 2: Week 12 | 35.8 |  |
  Participant 2: Week 48: number analyzed (Participants) | 1 | 0 | 0
  Participant 2: Week 48 | 39.6 |  |
  Participant 3: Baseline: number analyzed (Participants) | 0 | 1 | 0
  Participant 3: Baseline |  | 25.1 |
  Participant 3: Week 12: number analyzed (Participants) | 0 | 1 | 0
  Participant 3: Week 12 |  | 4.15 |
  Participant 3: Week 48: number analyzed (Participants) | 0 | 1 | 0
  Participant 3: Week 48 |  | NA — The 4-MU concentration at this time point was below the limit of quantitation |
  Participant 4: Baseline: number analyzed (Participants) | 0 | 1 | 0
  Participant 4: Baseline |  | 6.39 |
  Participant 4: Week 12: number analyzed (Participants) | 0 | 1 | 0
  Participant 4: Week 12 |  | 18.4 |
  Participant 4: Week 48: number analyzed (Participants) | 0 | 1 | 0
  Participant 4: Week 48 |  | 16.1 |
  Participant 5: Baseline: number analyzed (Participants) | 0 | 1 | 0
  Participant 5: Baseline |  | 17.3 |
  Participant 5: Week 12: number analyzed (Participants) | 0 | 1 | 0
  Participant 5: Week 12 |  | 5.85 |
  Participant 5: Week 48: number analyzed (Participants) | 0 | 1 | 0
  Participant 5: Week 48 |  | 22.2 |
  Participant 6: Baseline: number analyzed (Participants) | 0 | 1 | 0
  Participant 6: Baseline |  | 24.6 |
  Participant 6: Week 12: number analyzed (Participants) | 0 | 1 | 0
  Participant 6: Week 12 |  | 12.6 |
  Participant 6: Week 48: number analyzed (Participants) | 0 | 1 | 0
  Participant 6: Week 48 |  | 46.5 |
  Participant 7: Baseline: number analyzed (Participants) | 0 | 0 | 1
  Participant 7: Baseline |  |  | 3.25
  Participant 7: Week 12: number analyzed (Participants) | 0 | 0 | 1
  Participant 7: Week 12 |  |  | 6.56
  Participant 7: Week 48: number analyzed (Participants) | 0 | 0 | 1
  Participant 7: Week 48 |  |  | 4.83
  Participant 8: Baseline: number analyzed (Participants) | 0 | 0 | 1
  Participant 8: Baseline |  |  | 14.7
  Participant 8: Week 12: number analyzed (Participants) | 0 | 0 | 1
  Participant 8: Week 12 |  |  | 23.3
  Participant 8: Week 48: number analyzed (Participants) | 0 | 0 | 1
  Participant 8: Week 48 |  |  | 29.2
  Participant 9: Baseline: number analyzed (Participants) | 0 | 0 | 1
  Participant 9: Baseline |  |  | 13.1
  Participant 9: Week 12: number analyzed (Participants) | 0 | 0 | 1
  Participant 9: Week 12 |  |  | 8.86
  Participant 9: Week 48: number analyzed (Participants) | 0 | 0 | 1
  Participant 9: Week 48 |  |  | 7.58

ADVERSE EVENTS:
Time Frame: Day 1 after dosing through Week 48 (end of extension period)
Arm/Group | Migalastat Low Dose 50 mg | Migalastat Middle Dose 150 mg | Migalastat High Dose 250 mg
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat Low Dose 50 mg (N=2) | Migalastat Middle Dose 150 mg (N=4) | Migalastat High Dose 250 mg (N=3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat Low Dose 50 mg (N=2) | Migalastat Middle Dose 150 mg (N=4) | Migalastat High Dose 250 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Bifascicular block (Cardiac disorders) | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Mitral valve calcification (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Fabry's disease (Congenital, familial and genetic disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bronchitis acute (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Atrial pressure increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Echocardiogram abnormal (Investigations) | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 1 | 1
Electrocardiogram PR shortened (Investigations) | 0 | 0 | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 | 1 | 0
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 0 | 1
QRS axis abnormal (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral Artery occlusion (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Gliosis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.